CLINICAL TRIAL: NCT03645447
Title: Using a Diagnostic Taste Test as a Surrogate Biomarker to Predict Drug Effectiveness in Patients With Depression (MDD)
Brief Title: The Taste-Mood Diagnostic Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ranvier Health Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ranvier BRS 2.1
Record Dates: First submitted 2018-07-18; First posted 2018-08-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Depression; Diagnostic aid; Taste
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Taste tests will be undertaken, in order to establish taste thresholds. Observation of changes in taste thresholds with change in mood following antidepressant treatment may help develop a diagnostic test for depression. The taste test will not assist diagnosis of depression for the group of participants in this study, so the primary purpose is not diagnostic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taste test (Experimental): Participants newly diagnosed with depression will be presented with a series of sugar solutions of 9 different concentrations in pseudo-random order. The threshold at which each participant reliably detects the sugar taste is determined before and after a first antidepressant. Mood Questionnaires will be used to determine whether a participant is clinically depressed at the time of the taste test and 6 to 8 weeks later.
  Interventions: Diagnostic Test: Taste test

INTERVENTIONS:
Diagnostic Test: Taste test — A pseudo-randomised series of taste solutions are presented to the participant for identification as sugar or water, in order to establish their taste threshold.

SUMMARY:
The study looks at whether a taste test device can be used as a diagnostic aid for depression. Taste tests will be carried out before and after first use of an antidepressant (prescribed by the patient's GP) and then again six to eight weeks later a further taste test will be conducted. The results of these tests will be assessed to see if they correlate with the outcome of validated mood questionnaires carried out at the first and second visits.

DETAILED DESCRIPTION:
Research shows a clear link between taste sensitivity and depression, based on chemistry shared by the tongue and the brain. (Heath, T.P., Melichar, J.M., Nutt, D.J., Donaldson L.F. (2006) Human taste thresholds are modulated by serotonin and noradrenaline). The aim of this study is to investigate the use of a taste test in the diagnosis of depression and to predict drug effectiveness.

A test is carried out before and after ingesting a probe drug (first prescribed antidepressant) to assess change in taste. Standard validated questionnaires are used to assess mood on the day the first antidepressant is ingested and then again six to eight weeks later.

The study is a single centre, open label study using the patient's prescribed antidepressant as a probe with the primary objective of building on previous results obtained in a pilot study which used paroxetine as the probe drug (whether or not this was the drug chosen for treatment). The study is powered to test 240 patients, with a provision built in to the protocol for an interim analysis after 120 patients.

Participants will be followed up after six to eight weeks of usual clinical care, by means of follow up questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of previously untreated Major Depressive Disorder (MDD) of at least 3 weeks duration or new or recurrent MDD untreated before this episode (patients who have previously received treatment for MDD must have stopped taking antidepressant medication at least six weeks prior to entering the trial);
* Patients requiring pharmaceutical intervention as a treatment for MDD;
* Not suffering from any significant other mental or physical illness, such as confirmed psychosis, or end of life care.
* Receiving stable medical therapy for 30 days or longer before screening assessments;
* Be willing and able to comply with all visits and study related procedures;
* Not infected with coronavirus or needing to self-isolate
* Understands the study requirements and the treatment procedures and is able to provide written informed consent.

Exclusion Criteria:

* Already on antidepressant medication;
* Known or suspected hypersensitivity or intolerance to any probes, or any of their excipients;
* Relevant history or presence upon clinical examination, of cardiac, ophthalmologic, gastro-intestinal, hepatic, or renal disease or other condition known to increase risk of side effects of the probe drugs. This exclusion criterion is determined by the Site Investigator;
* Have a history or presence of neurological or confounding psychiatric conditions (such as stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, or schizophrenia),
* Patients with a diagnosis of chronic pain.
* Participation in another trial concurrently or within 30 days preceding enrolment that is deemed to interfere with this trial;
* Patients who are pregnant, or who are likely to become pregnant, will be excluded from the trial, as will breastfeeding mothers;
* Patients using supplements containing psychoactive herbs (for example St Johns Wort or 5-HTP (5-Hydroxytryptophan, also known as oxitriptan);
* Patients regularly using psychoactive stimulants and recreational drugs (for example MDMA (ecstasy/ methyl enedioxy methamphetamine), amphetamine, LSD (lysergic acid diethylamide), cocaine);
* Patients infected with coronavirus, or who are advised to self-isolate
* Patients who are unable or unwilling to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in taste threshold with antidepressant treatment | 6 weeks (per participant)
  Change in taste threshold between baseline and after ingestion of probe antidepressant
Change in mood (assessed by score on the Beck Depression Inventory) with antidepressant treatment | 6 weeks (per participant)
  Change in mood (assessed by score on the Beck Depression Inventory (BDI)) with antidepressant treatment is assessed. BDI scores may range from 0-63, where 0 demonstrates the lowest depression score and 63 the most severe depression.

SECONDARY OUTCOMES:
Change in mood with antidepressant treatment, measured by the Patient Health Questionnaire 9 (PHQ9) | 6 weeks (per participant)
  Change in mood with antidepressant treatment, measured by the Patient Health Questionnaire 9 (PHQ9). PHQ9 scores range from 0-27, where 0 is the score for the least depressed patients and 27 the most severely depressed patients.
Change in mood with antidepressant treatment, measured by the Generalised Anxiety Disorder 7 (GAD 7) Questionnaire | 6 weeks (per participant)
  Change in mood with antidepressant treatment, measured by the GAD 7 Questionnaire GAD 7 scores range from 0-21, where 0 is the score for the least anxious patients and 21 the most severely anxious patients.
User assessment of ease of use of the device and testing process. | 6 weeks (per participant)
  User views on ease of the testing process will be collected. Users will be asked to give ease of use a score from 1-5, where 1 is very easy and 5 is very difficult. Participants will also be asked whether they would use the taste test again.

CONTACTS AND LOCATIONS:
Overall Officials: David Adams, BDS, MSc, Principal Investigator — Ranvier Health Ltd
Locations (4):
- United Kingdom (4):
  - Jhoots Pharmacy, Bristol, Avon
  - Honiton Surgery, Honiton, Devon
  - Humber Teaching NHS Foundation Trust, Hull, Yorkshire
  - West Walk Surgery, Yate, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heath TP, Melichar JK, Nutt DJ, Donaldson LF. Human taste thresholds are modulated by serotonin and noradrenaline. J Neurosci. 2006 Dec 6;26(49):12664-71. doi: 10.1523/JNEUROSCI.3459-06.2006. PMID 17151269